CLINICAL TRIAL: NCT05267743
Title: A Multicenter, Double-blind, Randomized, Active-controlled Phase 4 Study to Evaluate the Efficacy and Safety of Tegoprazan in Patients With Erosive Reflux Disease
Brief Title: Study to Confirm the Safety and Efficacy of Tegoprazan in Patients With Healed Erosive Reflux Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: HK inno.N Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IN_APA_402
Record Dates: First submitted 2021-07-06; First posted 2022-03-04 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2022-07

CONDITIONS: Erosive Reflux Disease
MeSH Terms: interventions — tegoprazan; Lansoprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tegoprazan 50mg QD (Experimental): Tegoprazan 50mg tablet, once daily, oral administration
  Interventions: Drug: Tegoprazan 50mg QD
- Lansoprazole 30mg QD (Active Comparator): Lansoprazole 30mg capsule, once dauly, oral administration
  Interventions: Drug: Lansoprazole 30mg QD

INTERVENTIONS:
Drug: Tegoprazan 50mg QD — Tegoprazan 50mg tablets will be orally administered, once daily, for up to 2 weeks or 4 weeks.
  Arms: Tegoprazan 50mg QD
Drug: Lansoprazole 30mg QD — Lansoprazole 30mg tablets will be orally administered, once daily, for up to 2 weeks or 4 weeks.
  Arms: Lansoprazole 30mg QD

SUMMARY:
This study is designed to evaluate the efficacy and safety of Tegoprazan 50mg, compared to Lansoprazole 30mg in patients with healed erosive reflux disease confirmed by endoscopy following oral administration once daily(QD) of 2 weeks or 4 weeks.

DETAILED DESCRIPTION:
This is a double blind, radomized, active-controlled, phase 4 study. Subjects will be randomly assigned to one of the two treatment groups (Tegoprazan 50mg, Lansoprazole 30mg)

ELIGIBILITY:
Inclusion Criteria:

1. Erosive eshophagitis(LA calssfication Grades A to D) with in 30 days prior to Randomization
2. Those who have experienced heartburn symptoms within 7 days prior to Visit 1(screening date)

Exclusion Criteria:

1. Unalbe to undergo upper GI endoscopy
2. H. pylori positive
3. Those who cannot write a clinical trial subject diary
4. Presence of esophageal stricture, ulcerated stricture, gastroesophageal varix, long segment Barrett's esophagus with >3cm length(LSBE), eosinophilic oesophagitis, active digestive ulcer or gastric bleeding on an upper GI endoscopy

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 218 (Actual)
Dates: Start 2021-02-16 (Actual); Primary Completion 2022-05-25 (Actual); Study Completion 2022-05-25 (Actual)

PRIMARY OUTCOMES:
4 weeks cumulative ERD healing rate(%) | 4 weeks
  Healing is defined as "not present" erosions or fissures according to the LA classification.

SECONDARY OUTCOMES:
2 weeks ERD healing rate(%) | 2 weeks
  Healing is defined as "not present" erosions or fissures according to the LA classification.
Healing rate(%) at 2 weeks and 4 weeks according to CYP2C19 genotype type | 2 weeks or 4 weeks
  Extensive Metaboliser (EM), Intermediate Metaboliser (IM), Poor Metaboliser (PM)
Percentage of days without heartburn through the clinical trial subject dairy (%) | 2 weeks or 4 weeks
  On days with no symptoms of heartburn, '0. It is defined as a case assessed as having no symptoms.
RDQ (Reflux Disease Questionnaire) evaluation(mean change in severity) | 2 weeks or 4 weeks
  Average scale change in RDQ severity and frequency at 2 weeks and 4 weeks after administration compared to before administration of investigational drugs for each category (heartburn, indigestion, acid reflux)
Incidence of Adverse Events [Safety] | 2 weeks or 4 weeks
  Physical examination(weight-kg)(height-cm), vital signs(SBP, DBP, heart rate, body temperature), adverse reactions, blood chemistry test

CONTACTS AND LOCATIONS:
Overall Officials: Suk Chae Choi, Principal Investigator — Wonkwang University Hospital
Locations (1):
- Wonkwang University Hospital, Iksan, Muwang-ro 895, South Korea

REFERENCES:
- [Derived] Shin CM, Choi SC, Cho JW, Kim SY, Lee OJ, Kim DH, Cho YK, Lee JY, Lee SK, Shin JE, Kim GH, Park SY, Hong SJ, Jung HK, Lee SJ, Youn YH, Jeon SW, Sung IK, Park MI, Lee OY. Comparison of Tegoprazan and Lansoprazole in Patients With Erosive Esophagitis up to 4 Weeks: A Multi-Center, Randomized, Double-Blind, Active-Comparator Phase 4 Trial. Neurogastroenterol Motil. 2025 Jan;37(1):e14969. doi: 10.1111/nmo.14969. Epub 2024 Nov 25. PMID 39587796